CLINICAL TRIAL: NCT04438343
Title: Effects of Impairment-Specific and Augmented Intervention on Turning Performance in Individuals With Chronic Stroke
Brief Title: Impairment-Specific and Augmented Intervention on Turning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM109070F
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Other: Impairment-specific and augmented intervention
- control group (Active Comparator)
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Impairment-specific and augmented intervention — Balance and lower extremities strength training
  Arms: experimental group
Other: Conventional physical therapy — Trunk and upper extremity training
  Arms: control group

SUMMARY:
The objective of this study is to investigate the effects of the impairment-specific and augmented intervention based balance and strength training on turning performance in individuals with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* ≧ 6 months post first-ever stroke with unilateral motor deficits
* ≧20 years of age
* The ability to walk independently for at least 7 m with or without using walking aids
* Score ≧ 24 of 30 on the Mini-Mental State Examination

Exclusion Criteria:

* Unstable medical conditions (e.g., deep vein thrombosis, aspiration pneumonia, or superimposed sepsis)
* History of other diseases known to interfere with participation in the study (e.g., heart failure, hemineglect, or diabetic neuropathy)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Turning performance | Change from baseline at 4 week
  Using a turning characteristic evaluation system to evaluate the swing time, stance time, turning speed, and stride length of the participants during turning

SECONDARY OUTCOMES:
Balance | Change from baseline at 4 week
  Berg Balance Scale Limits of stability (LOS) using NeuroCom Smart Balance Master (NeuroCom International, Clackamas, OR)
Strength | Change from baseline at 4 week
  Using handheld dynamometer
Straight walking performance | Change from baseline at 4 week
  Using GAITRite system (CIR system, Inc, Havertown, PS) calculate walking speed, cadence, swing time, stance time, and step length
Timed up and go test | Change from baseline at 4 week
Falls Efficacy Scale International (Chinese) | Change from baseline at 4 week
Stroke Impact Scale (SIS) Taiwan version | Change from baseline at 4 week

CONTACTS AND LOCATIONS:
Locations (1):
- Yea-Ru Yang, Taipei, Beitou, Taiwan